CLINICAL TRIAL: NCT05319977
Title: Mobile Behavioral Intervention to Reduce Maternal Drinking in South Africa
Brief Title: Maternal Alcohol Reduction Intervention in South Africa [MaRISA]
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Medical Research Council, South Africa (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Yukiko Washio, Senior Research Psychologist, RTI International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0217974; R21AA029048 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-04-11 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Maternal; Alcohol Use, Affecting Fetus
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile incentive-based intervention (Experimental): Contingent incentives on abstinence from alcohol; Text-based health promotion support
  Interventions: Behavioral: Mobile incentive-based intervention

INTERVENTIONS:
Behavioral: Mobile incentive-based intervention — a technology-based behavioral intervention to address maternal alcohol use with mobile breathalyzer technology or/and urinalysis for biochemical verification of alcohol use, contingent financial incentives on alcohol abstinence, and text-based health promotion.

SUMMARY:
This application proposes to develop and test a technology-based behavioral intervention to address maternal alcohol use in South Africa (SA). SA reports the highest per capita rates of alcohol consumption in the world and has one of the world's highest rates of lifelong disorders called fetal alcohol spectrum disorders (FASD). Prenatal alcohol use is often associated with exposure to gender-based violence, and an increase in gender-based violence due to the uncertainty and economic impact of COVID-19 is of a major concern. Recent evidence also showed that alcohol use during lactation significantly compromises child development in children exposed to alcohol through breastfeeding, and the adverse effect of postpartum alcohol use while breastfeeding was independent of prenatal alcohol exposure. Average breastfeeding duration in SA is beyond 1 year, and over 40% of mothers with and without a history of prenatal drinking report alcohol use while breastfeeding. A community-based behavioral intervention involving case management helps reduce prenatal alcohol use but is labor intensive, challenging the feasibility of widespread implementation in economically disadvantaged communities especially during the COVID-19 pandemic with limited social contact. An efficacious behavioral intervention to reduce alcohol use during pregnancy and lactation needs to be developed that is acceptable and feasible in economically disadvantaged communities, for women with transportation difficulties, or during the COVID-19 pandemic with limited social contact. The proposed intervention will incorporate mobile breathalyzer technology, contingent financial incentives, and text-based health promotion and referrals on gender-based violence, maternal infant health, and psychosocial issues including the impact of COVID-19 in the context of maternal alcohol use. Specific aims are (1) to develop and pretest a technology-based behavioral intervention to help women abstain from alcohol use during pregnancy and lactation via formative qualitative research with women who are pregnant or breastfeeding with a recent history of alcohol use, clinic and community stakeholders, and an established Community Collaborative Board in Cape Metropole, SA, and (2) to examine the acceptability and feasibility of the intervention on alcohol use during pregnancy and lactation by pilot testing the mobile technology-based platform with 60 women who are pregnant or postpartum. Acceptability will be assessed at follow-ups, and feasibility will include recruitment capability, process measures, and intervention outcomes. With the evidence of acceptability and feasibility of the proposed intervention, a large randomized clinical trial will become essential to establish efficacy of the intervention. The potential settings that can remotely incorporate the proposed behavioral intervention include primary care clinics, substance use treatment programs, and publicly funded programs for maternal/infant populations in SA, the United States, and other countries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant (≤28 ges wks) or postpartum (≤3 mos)
* Have reported alcohol use during the current pregnancy or lactation
* Positive for alcohol use by urinalysis
* Have their own mobile phone
* Intend to breastfeed for 6 months
* Voluntarily consent

Exclusion Criteria:

* Participated in focus group discussions or pretesting will not be eligible for pilot testing
* Serious medical problems threatening their current pregnancy or current suicidal thoughts or attempts in the past month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South African Medical Research Council, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After the main findings are published, we welcome other researchers who want to analyze the data in other ways.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Erasmus-Claassen LA, Mpisane N, Petersen Williams P, Browne FA, Myers B, Wechsberg WM, Parry CDH, Taylor SN, Washio Y. Participant experiences with a text message and contingency management intervention for alcohol use during pregnancy and lactation in Cape Town, South Africa. Addict Sci Clin Pract. 2025 Jul 29;20(1):59. doi: 10.1186/s13722-025-00594-7. PMID 40734177

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Incentive-based Intervention
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 54
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Mixed | 46
  Race/Ethnicity: Black | 14
Region of Enrollment [Number; unit: participants]
  South Africa | 60

OUTCOME MEASURES:

1. Primary Outcome: Urine Ethylglucuronide (EtG) Testing
Description: Number and proportion of participants who were tested negative of alcohol use in urine samples.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 60
Participants | 0

2. Primary Outcome: Urine Ethylglucuronide (EtG) Testing
Description: Number and proportion of participants who were tested negative of alcohol use in urine samples.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 57
Participants | 31

3. Primary Outcome: Urine Ethylglucuronide (EtG) Testing
Description: Number and proportion of participants who were tested negative of alcohol use in urine samples.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 52
Participants | 31

4. Primary Outcome: Self-reported Recent Drinking With Timeline Followback
Description: Self-reported use of daily alcohol by the number of standard drinks based on the definition in South Africa (e.g., 12 g per standard drink). The minimum value is 0 and the maximum has no limit in value. The higher the score is, the worse the outcome would be.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: the number of standard drinks per day
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 60
the number of standard drinks per day | 9 (5.6)

5. Primary Outcome: Self-reported Recent Drinking With Timeline Followback
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: the number of standard drinks per day
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 57
the number of standard drinks per day | 3 (5.4)

6. Primary Outcome: Self-reported Recent Drinking With Timeline Followback
Description: as for outcome 4
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: the number of standard drinks per day
Arm/Group | Mobile Incentive-based Intervention
Number analyzed (Participants) | 52
the number of standard drinks per day | 2 (4.9)

ADVERSE EVENTS:
Time Frame: 3 months per participant
Arm/Group | Mobile Incentive-based Intervention
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 5/60
Other Adverse Events (participants affected / at risk) | 2/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile Incentive-based Intervention (N=60)
neonatal death (Pregnancy, puerperium and perinatal conditions) | 1 — Neonatal death occurred, and counseling was offered to the participant.
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile Incentive-based Intervention (N=60)
Intoxication (Psychiatric disorders) | 1
Abscesses on breasts (Pregnancy, puerperium and perinatal conditions) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT05319977/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT05319977/SAP_001.pdf
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT05319977/ICF_002.pdf